CLINICAL TRIAL: NCT04591574
Title: Anaemia Management With Red Blood Cell Transfusion to Improve Post-intensive Care Disability: a Randomised Controlled Trial (The ABC Post-intensive Care Trial)
Brief Title: ABC - A Post Intensive Care Anaemia Management Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC19089
Record Dates: First submitted 2020-09-03; First posted 2020-10-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Anemia Acute; Fatigue; Physical Disability; Quality of Life
Keywords: Post Intensive Care Recovery; Blood Transfusion; Physical Function; Moderate-Severe Anaemia; Systemic Inflammation; Impaired Erythrogenesis
MeSH Terms: conditions — Fatigue | interventions — Erythrocyte Count; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): All patients will receive a single unit red blood cell (RBC) transfusion post randomisation. Single RBC transfusions will subsequently be administered to achieve and maintain haemoglobin (Hb) concentration of 100-120g/L unitl hospital discharge. Hb measured at least weekly in hospital.
  Interventions: Biological: Red Blood Cells (Transfusion)
- Usual care group (Active Comparator): Current usual care transfusion practice, namely single RBC transfusions when Hb 70g/L or less (or modified according to clinician decision) to achieve target Hb 70-90g/L. HB measured at least weekly in hospital
  Interventions: Biological: Red Blood Cells (Transfusion)

INTERVENTIONS:
Biological: Red Blood Cells (Transfusion) — Participants will receive RBC transfusions in accordance with trial protocol (intervention group) or usual care, which is in accordance with the NICE guidelines

SUMMARY:
On discharge from intensive care (ICU) patients are often severely anaemic (have a low level of haemoglobin (Hb) in their red blood cells (RBC)). Anaemia can persist for many months making patients feel tired and fatigued. Regaining pre-illness health and energy levels can take a long time.

The ABC Post Intensive Care Trial will be the first trial to investigate if an anaemic ICU patient's health can be improved by treating with RBC transfusions following ICU discharge. We will compare the current approach as per national guidelines (restrictive transfusion), with a more active transfusion regime to correct anaemia from ICU discharge to hospital discharge.

The trial will take place in acute hospitals throughout the UK where patients are discharged after a period of time in ICU.

Patients discharged, or ready for discharge from ICU will be approached to consider participation in the trial. Once Hb level drops below 94g/L they would become eligible for inclusion (subject to meeting inclusion/exclusion criteria). The main indication for being excluded from participating in the trial is that transfusions are contraindicated (not appropriate for the patient) or they have an objection to blood transfusions.

Group allocation will be randomly assigned at ICU discharge. We will explore which patients benefit most from transfusions and those who gain no benefit.

Patients will have their Hb level checked at least weekly whilst in hospital and based on the result will have RBC transfusions as required according to the treatment regime they were randomised to.

Part of the research is based on self-reported quality of life so participants will be asked to complete a number of questionnaires at set time-points from randomisation to 6 months post randomisation.

Each participant will be actively on trial for approximately 6 months. The five-year follow will be done using routinely collected data from national databases.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received level 3 ICU care at any time point during the current hospital admission (defined as advance respiratory support and/or at least two organ support).
* Patient considered ready for discharge from ICU by the caring clinical team.
* Hb less than or equal to 94g/L when ready for ICU discharge or during the first seven days following the decision by the treating clinician that the patient is ready for ICU discharge.
* 16years of age or older
* Patient expected to remain in study hospital until hospital discharge.
* Consent provided (by participant or in accordance with appropriate mental capacity legislation for the site).

Exclusion Criteria:

* Contraindication or objection to RBC transfusion
* Active bleeding when screened
* Primary neurological ICU admission diagnosis
* Patients discharged from the ICU following cardiac surgery
* Currently receiving or planned to receive end-of-life care
* Not expected by clinical team to survive to hospital discharge
* Patient with a proven chronic haematological disease that requires regular RBC transfusion to treat anaemia
* Patient with dialysis-dependent chronic renal failure prior to ICU admission
* Patient receiving regular erythropoietin (or any erythropoiesis stimulating agent) treatment for anaemia prior to ICU admission
* Unable to obtain consent (frompatietn or in accordance with appropriate mental capacity legislation for the site)
* Readmission to ICU during current hospitalisation episode and not enrolled following previous ICU admissions
* Patient recovering following liver transplantation, kidney transplantation, or combined kidney/pancreas transplantation
* Patient recovering from variceal bleeding due to chronic liver disease
* Prisoners
* Patient due for imminent hospital discharge within the next 24 hours

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Physical component score (PCS) of the SF-36 Health Related Quality of Life (HRQoL) questionnaire at 3 months post randomisation | 3 months post randomisation

SECONDARY OUTCOMES:
PCS of the SF-36 HRQoL questionnaire (and its four sub-domains) at 1 and 6 months post randomisation. | 6 months post randomisation
Patient Fatigue (Fatigue Severity Scale (FSS)) at 1, 3 and 6 months post randomisation | 6 months post randomisation
Mental Component Score of SF-36 (and its four sub-domains) at 1, 3 and 6 months post randomisation | 6 months post randomisation
Activities of Daily Living (ADLs) (from WHODAS questionnaire) at 3 months post randomisation | 3 months post randomisation
Patients alive at 1, 3, and 6 months post-randomisation | 6 months post randomisation
Patients alive at 5 years post-randomisation derived from data linkage | 5 years post randomisation
Haemoglobin concentration at 1 month post-randomisation | 1 month post randomisation
Post-ICU length of hospital stay | Variable according to patient's length of hospital stay
Care costs during 6 months post-randomisation | 6 months post randomisation
Incremental cost per QALY at 6 months | 6 months post randomisation
Care costs derived from data linkage during 5 years post-randomisation | 5 years post randomisation
Protocol compliance (during intervention index hospital stay) | Throughout the study, for an average of 1 month
  Proportion of participants compliant with the study intervention as per protocol (%).
Hb concentration (during index hospital stay) | Throughout the study, for an average of 1 month
RBC use (during 3 months follow up) | 3 months post randomisation
New Infections (during 3 months follow-up) | 3 months post randomisation
Transfusion-related adverse events (during 3 months follow-up) | 3 months post randomisation
Major adverse cardiovascular events (MACE; during 3 months follow-up) | 3 months post randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Walsh TS, Emerson L, Singleton J, Locherty R, Hope D, Cholbi S, Giddings A, Macdonald A, Lone N, Docherty AB, Mead G, Stanworth SJ, Drakesmith A, Roy NBA, Hall P, Neilson AR, Pollock R, Rodriguez A, Norrie J, Weir CJ, Shah A, Griffith D. Anaemia management with red blood cell transfusion to improve post-intensive care disability: Protocol for the ABC post-ICU randomised controlled trial. J Intensive Care Soc. 2025 Nov 12:17511437251374884. doi: 10.1177/17511437251374884. Online ahead of print. PMID 41244217
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066